CLINICAL TRIAL: NCT06807853
Title: SYMPTOM-ACCESSMENT in SUBJECTS with AXIAL SPONDYLOARTHRITIS with PATIENT-REPORTED OUTCOMES and MOBILITY TRACKING with SMARTWATCHES VIA SPECIALLY PROGRAMMED STUDY-APP to EVALUATE the EFFICACY of MOVEMENT and IMPLEMENT CONCRETE MOVEMENT RECOMMENDATIONS
Brief Title: A LONGITUDINAL OBSERVATIONAL STUDY to EVALUATE the EFFICACY of MOVEMENT and IMPLEMENT CONCRETE MOVEMENT RECOMMENDATIONS with the HELP of MOBILITY TRACKING with SMARTWATCHES in SUBJECTS with AXIAL SPONDYLOARTHRITIS
Acronym: SPARTAKUS
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Collaborators: Novartis (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Valentin Schäfer, Prof. Dr., University Hospital, Bonn
Other Study IDs: 115/23; MAIN457A_FVMBO009 (Other: Novartis)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Axial Spondyloarthritis; Axial Spondyloarthritis (AxSpA); Axial Spondylarthritis (r-axSpA); Axial Spondyloarthopathy; Axial Spondyloarthritis and Ankylosing Spondylitis; Axial Spondyloarthritis, Non-Radiographic; Axial and Peripheral Spondyloarthritis
Keywords: Mobility Tracking; Patient-Reported Outcomes (PROs); Disease Activity; Smartwatch; Study-App; Mobile Device; Movement Recommedations
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Smartwatch — Smartwatch AppleWatch SE to track Mobility

SUMMARY:
Axial spondyloarthritis (axSpa) is a chronic inflammatoric autoimmune disease of the back with a prevalence around 1,4% (1) . In patients decreased function and decreased quality of life as well as chronic pain are strong burdens . Despite modern treatments like biological agents just 25% of the patients are at remission (2) . Besides the pharmacological treatment physical activity is known to be very important to gain disease control. A low physical activity is related to a higher disease activity and a high physical activity to better disease control. Until now there is no structured capture of the daily movements of patients with axial spondylarthritis in clinical practice. Our goal is to analyse the relationship between movement and disease activity and to implement concrete recommendations for movement in patients with axSpa.

The primary objective of the study is to investigate which type, frequency and intensity of movement are helpful in gaining and remaining disease control in patients with axSpa.

Methods This monocentric longitudinal study recordes movement, sport and physical parameters like heart frequency and heart rate variability through an observational period of 6 month via smartwatch. Meanwhile we record disease activity, pain and functional outcomes with regular surveys every two weeks. Patients in every phase of disease are eligible for inclusion, but they do must have an own iPhone due to software reasons. Data is collected in a specially programmed study-app. Fifty participants will be included in this study. Until now we have 24 patients included since april 2024. Patients come to clinic every 3 month as this is our standard in outclinic patients. We than do anamnesis and a physical examination. After the study period of 6 month we transmit the mobility and disease-related data of the surveys of the patients mobile device to our system.

The primary endpoint is to find exact recommendations for concrete movement in patients with axSpa.

So this is the first study that wants to give concrete recommendations for movement in patients with axSpa with the help of mobility tracking with smartwatches. This could help to prevent flares and also to recover quicker from a flare.

1. López-Medina und Moltó, "Update on the epidemiology, risk factors, and disease outcomes of axial spondyloarthritis".
2. Pina Vegas u. a., "Factors associated with remission at 5-year follow-up in recent-onset axial spondyloarthritis: results from the DESIR cohort".

ELIGIBILITY:
Inclusion Criteria:

* Patients with Axial Spondyloarthritis
* Patients do must have an own iPhone due to software reasons
* do must be willing and able to wear a Smartwatch
* do must be able to regularly fill out the PROs at home

Exclusion Criteria:

* no iphone
* no physical or mental Ability to wear a Smartwatch
* no physical or mental Ability to regularly fill out the PROs at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prensenting in University Clinic Bonn, Department of Rheumatology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Recommendation for Rate of steps per day | From enrollment to Week 24
  values: 0- >20.000
Recommendation for minutes of training per day | From enrollment to Week 24
Recommendation for minutes of standing per day | From enrollment to Week 24
Recommendation for average heart frequence per day | From enrollment to Week 24
Recommendation for heart rate variability | From enrollment to Week 24

SECONDARY OUTCOMES:
Numeric rating scale pain at week 24 | From enrollment to Week 24
  minimum value: 0 maximum value: 10, higher scores mean a worse outcome.
Disease Activity depending on Movement of Patient | From enrollment to Week 24
  using:
  * Numeric rating scale disease activity (NRS DA, values 0-10, best value: 0, worst value: 10),
  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI, values 0-10, best value 0, worst value 10);
  * Bath Ankylosing Spondylitis Functional Index (BASFI, values 0-10, best value 0, worst value 10),
  * Gesundheitsindex Axiale Spondyloarthritis - ASA-Score (ASAS, values: 0-17, best value: 0, worst value: 17),
  * European Quality of Life 5 Dimensions Score (EQ-5D, for each dimension a 1-digit number expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, best combined value 11111, worst combined value 55555),
  * Morning stiffness Score (scale from 0 minutes to >60 minues, worst value:>60 min),
  * Facit Fatigue Score (values 8-44, best value 44, value < 30: suspicious for severe fatigue),
  * Funktionsfragebogen Hannover (FFbH, values 0- 36, best value: 36, worst value 0 )

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Department for Rheumatology, Bonn, North Rhine-Westphalia, Germany